CLINICAL TRIAL: NCT06556017
Title: Assessing the Efficacy of ChatGPT in Detecting Surgical Site Infections Following Elective Colorectal Surgery
Brief Title: Assessment of the Efficacy of ChatGPT in Detecting Surgical Site Infections Following Elective Colorectal Surgery
Acronym: ChatCCR
Status: Completed | Type: Observational
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep M Badia, Prof, Hospital de Granollers
Other Study IDs: HGG2024_03
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Surgical Site Infection
Keywords: Surgical Site Infection; Surveillance; Artificial intelligence; ChatGPT; natural language processing
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients assessed for ILQ using the standard manual surveillance method: Patients undergoing colorectal surgery enrolled in the nationwide ILQ surveillance programme and assessed for ILQ using the standard manual surveillance method.
  Interventions: Diagnostic Test: Diagnosis of SSI
- ILQ patients assessed by Open IA's ChatGPT 4 chatbot: Patients undergoing colorectal surgery enrolled in the nationwide ILQ surveillance programme and assessed for ILQ using the Open IA's ChatGPT 4 chatbot.
  Interventions: Diagnostic Test: Diagnosis of SSI

INTERVENTIONS:
Diagnostic Test: Diagnosis of SSI — Comparison of the manual system and ChatGPT for SSI diagnosis in colorectal surgery procedures enrolled in the SSI surveillance programme.

SUMMARY:
Epidemiological surveillance is one of the eight core components of the World Health Organization Infection Prevention and Control Programmes. These include surveillance programmes for surgical site infection (SSI).

At present, for SSI surveillance, infection control teams perform a manual time-consuming work, which could make a transition to automated surveillance leveraging the new information technology.

This study aimed to evaluate the ability of ChatGPT-4o to detect surgical site infection at the three anatomical levels.

DETAILED DESCRIPTION:
Healthcare-associated infections (HAIs) have a negative impact on patient health, represent a significant healthcare and economic burden on healthcare systems and are considered the most preventable cause of serious adverse events in hospitalised patients.

Epidemiological surveillance is one of the eight core components of the World Health Organization (WHO) Infection Prevention and Control Programmes. These include surveillance programmes for surgical site infection (SSI), which have proven to be effective in all types of surgery and in a variety of settings.

For a programme to be effective, surveillance for HCAIs must be active, prospective and continuous, comprising a surveillance period up to 30-90 days post-intervention, to cover the high rate of SSIs detected after discharge.

At present, infection control teams perform a manual, prospective, time-consuming and almost artisanal work, which should make a transition to automated or semi-automated surveillance that leverages the possibilities offered by today's information technology.

The evolution of surveillance systems should benefit from this new possibilities offered by artificial intelligence, allowing automated detection of suspected SSI adverse events from clinical course text, microbiology reports or coding of diagnoses, procedures, complications and readmissions.

This pilot study aims to evaluate the ability of ChatGPT to detect surgical site infections (SSI) at the three anatomical levels described by the CDC. The aim is to retrospectively compare the results of the AI chatbot in diagnosing SSI, trained using the US CDC definition criteria, with a cohort of elective colorectal surgery patients evaluated through a nationwide nosocomial infection surveillance system.

ELIGIBILITY:
Inclusion Criteria:

* Elective colorectal resection

Exclusion Criteria:

* Emergency surgery
* Infection present at operation
* Previous intestinal stoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective colorectal surgery in Catalonia in the period 2020-2022
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of surgical site infection | 30 days
  Rate of Surgical site infection according to the definitions of the CDC-NHSN (Centers for Disease Control and Prevention-National Healthcare Safety Network)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Badia JM, Casanova-Portoles D, Membrilla E, Rubies C, Pujol M, Sancho J. Evaluation of ChatGPT-4 for the detection of surgical site infections from electronic health records after colorectal surgery: A pilot diagnostic accuracy study. J Infect Public Health. 2025 Feb;18(2):102627. doi: 10.1016/j.jiph.2024.102627. Epub 2024 Dec 18. PMID 39740340